CLINICAL TRIAL: NCT04631497
Title: Assessment of Stress, Depression and Anxiety in Healthcare Caring for Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, Ph.D. M.D., Jagiellonian University
Other Study IDs: 1072.6120.161.2020
Record Dates: First submitted 2020-11-09; First posted 2020-11-17 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Depression
Keywords: Healthcare Workers; COVID-19; Mental Health Outcomes
MeSH Terms: conditions — Depression; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare workers: The study will cover employees of the Intensive Care Unit - nurses and doctors working with patients with COVID-19 infection. Test takers will be over the age of 18 and under the age of 70, female and male.
  Interventions: Diagnostic Test: test

INTERVENTIONS:
Diagnostic Test: test — 1. Beck's Test
  2. Test STAI
  3. Test PSS
  4. the scale of the fascination with death
  5. COPE

SUMMARY:
Medical personnel working in the Intensive Care Unit will be examined by means of tests. Their aim is to check how work-related stress in a potentially lethal threat affects the occurrence of depression, stress, anxiety and sleep disorders. We also want to check whether people working in such extremely difficult conditions show no greater interest in death.

DETAILED DESCRIPTION:
Every day medical staff working in very difficult conditions of intensive care. The COVID-19 virus outbreak has set another difficult task for doctors and nurses who have previously had a lot of contact with the death of their patients. The appearance of the COVID-19 virus and, above all, the inability to effectively treat the infection causes an additional psychological stimulus in medical personnel.

The aim of the study is to assess the occurrence of psychiatric disorders in medical personnel dealing with patients suffering from COVID-19 using various psychological tests.

ELIGIBILITY:
Inclusion Criteria:

adult employees of the Intensive Care Unit, agreeing to undergo the tests.

Exclusion Criteria:

* patient's refusal to participate in the study
* not understanding the test questions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University Hospital in Cracow ICU depratment
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Depression | 1 month
  Beck's test the BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used differ from the original:
  0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression
Stress | 1 month
  Perceived Stress Scale (PSS)
  The PSS predicts both objective biological markers of stress and increased risk for disease among persons with higher perceived stress levels. For example, those with higher scores (suggestive of chronic stress) on the PSS fend worse on biological markers of aging, cortisol levels, immune markers, depression, infectious disease,wound healing, and prostate-specific antigen levels in men. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positivelystated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 item scale can be made fromquestions 2, 4, 5 and 10 of the PSS 10 item scale.
Deal with Stress | 1 month
  COPE test It is a self-written tool consisting of 60 statements, to which the respondent responds on a 4-point scale. It allows the assessment of 15 strategies for responding to stressful situations.

SECONDARY OUTCOMES:
Stress 2 | 1 month
  the scale of the fascination with death The Death Obsession Scale (DOS) was made by Abdel-Khalek. It was intended to be a main component in the death distress const.ruct: death anxiety, death depression, and death obsession. The DOS assesses a multidimensional trait. It is responded to on a five-point Likert-type rating scale as follows: No (1), A little (2), A fair amount (3), Much (4) and Very much (5). The total score can range from 15 to 75.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Skladzien, Ph.D. M.D., Principal Investigator — Jagiellonian University
Locations (1):
- University Hospital in Cracow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided